CLINICAL TRIAL: NCT05997186
Title: Sensory Recovery and Functional Outcome After Reinnervated Profunda Artery Perforator Flap for Oral Cavity and Oropharyngeal Defect Reconstruction - Prospective Pilot Study
Brief Title: Reinnervated PAP Flap for Oral Cavity and Oropharyngeal Defect Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-00938; mu23schaefer
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Oral Cavity Defect; Oropharynx Defect
Keywords: reconstruction with a free reinnervated profunda artery perforator flap; sensory recovery

STUDY DESIGN:
Intervention Model Description: Prospective case series (pilot study)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgery (Other): Oral cavity and oropharyngeal defect reconstruction
  Interventions: Procedure: Surgical reconstruction

INTERVENTIONS:
Procedure: Surgical reconstruction — Surgical reconstruction with a free reinnervated profunda artery perforator flap

SUMMARY:
The aim of this study is to investigate sensory recovery and functional outcomes following oral cavity and oropharyngeal defect reconstruction with reinnervated PAP (profunda artery perforator) flaps.

DETAILED DESCRIPTION:
Tumor resections involving the oral cavity or oropharynx cause significant functional deficits in swallowing and speech and subsequently impair the patients' quality of life. The anterolateral thigh (ALT) flap is widely regarded as a workhorse flap to reconstruct such defects. Previous studies assessing recovery of reinnervated ALT flaps reported superior sensory recovery, improved swallow function, and improved overall patient satisfaction in patients with reinnervated flaps compared with patients who received ALT flap reconstruction without sensory reinnervation. Recently, the profunda artery perforator (PAP) flap has been proposed as an alternative donor site in malnourished patients with thin lateral thigh thickness. However, reinnervation of PAP flaps has not been described. The study assesses sensory recovery after defect reconstruction with the reinnervated profunda artery perforator flap using already approved, non-invasive testing (Semmes-Weinstein monofilament testing, two-point discrimination, temperature, pain perception)

ELIGIBILITY:
Inclusion Criteria:

- Patient with defect involving the oral cavity or oropharynx who undergo reconstruction with a free reinnervated profunda artery perforator flap

Exclusion Criteria:

* <18 years old
* Defect localizations other than the oral cavity or oropharynx
* Not able to give informed consent
* Inability to follow the procedures of the study, e.g., due to psychological disorders, dementia
* Inability or contraindications to undergo the investigated intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Change in Semmes-Weinstein monofilament testing | before surgery and 3, 6 and 12 month after surgery
  The Semmes-Weinstein Monofilament test is a sensory assessment tool. This assessment tool consists of a set of monofilaments that vary in thickness and diameter, the gradient forces of these monofilaments ranges from .086 gm to 448gm. These monofilaments are used to map out sensory loss or recovery.
  Semmes-Weinstein monofilament testing will be performed at the tip (distal 1 cm) and the dorsum of the reconstructed flap/neo-tongue. Semmes-Weinstein monofilament testing will also be performed in the profunda artery perforator flap territory on the ipsilateral and contralateral thigh. For this purpose, the investigators will use the "Baseline FoldUp Monofilament Evaluator Set with Case".
Change in two-point discrimination test | before surgery and 3, 6 and 12 month after surgery
  The two-point discrimination test is used to assess if the patient is able to identify two close points on a small area of skin, and how fine the ability to discriminate this are. It will be measured using "Dellon Disk Criminator"
Change in temperature perception | before surgery and 3, 6 and 12 month after surgery
  Hot (50 degrees Celsius) and cold (4 degrees Celsius) temperature perception will be assessed by use of a small test tube filled with water at the appropriate temperatures.
Change in pain perception | before surgery and 3, 6 and 12 month after surgery
  Pain perception will be assessed with a 27-gauge needle.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole E. Speck, Dr. med., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Speck NE, Haumer A, Pfister P, Muller L, Gahl B, Burger M, Largo RD, Schaefer DJ, Ismail T. Neurotized profunda artery perforator flap for subtotal tongue reconstruction - Prospective case series. J Plast Reconstr Aesthet Surg. 2024 Aug;95:35-42. doi: 10.1016/j.bjps.2024.05.028. Epub 2024 May 31. PMID 38875869